CLINICAL TRIAL: NCT06457516
Title: Comparison the Effectiveness of Mirror Therapy VS Music Therapy for Balance and Gait Training in Post Stroke Hemiplegic Patients: Randomized Control Trial
Brief Title: Comparison the Effectiveness of Mirror Therapy VS Music Therapy for Training in Post Stroke Hemiplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/550
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Mirror Movement Therapy; Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy (Experimental)
  Interventions: Combination Product: Mirror Therapy
- Music Therapy (Other)
  Interventions: Other: Music Therapy

INTERVENTIONS:
Combination Product: Mirror Therapy — A mirror is used to create a reflective illusion of an affected limb in order to trick the brain into thinking movement has occurred without pain, or to create positive visual feedback of a limb movement. It involves placing the affected limb behind a mirror.
  Arms: Mirror Therapy
Other: Music Therapy — Music therapy, an allied health profession, the clinical and evidence-based use of music interventions to accomplish individualized goals
  Arms: Music Therapy

SUMMARY:
A randomized clinical trial was performed on hemiplegic post-stroke patients with a sample size of 50 (25 in each group).

DETAILED DESCRIPTION:
It was a single-blinded study. Mirror therapy was given to group A and music therapy was given to group B. Our findings support the alternate hypothesis. This indicates the small effect size for BBS in group A and the moderate effect size for the gait assessment scale in favor of group A.

ELIGIBILITY:
Inclusion Criteria:

* ischemic and hemorrhagic post stroke hemiplegic patients
* patients of age 40-60 years
* no visual perception dysfunction

Exclusion Criteria:

* patients with fracture of upper or lower limb
* patient with comorbidities
* patients with hearing issues
* patients with cognitive disabilities
* patient with other neurological disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
BBS (berg balance scale) | 6 Month
  A score of 56 indicates functional balance. A score of < 45 indicates individuals may be at greater risk of falling. A score of ≤49 indicates a risk of falls in individuals with stroke.
FGA (functional gait assessment scale) | 6 Months
  The normal score on the FGA would be considered >27/30; for adults from ages 60 to 80 years, the normal score on the FGA would be considered >24/30; and for adults over the age of 80 years, the normal score would be considered >19/30

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudhary Muhammad Akram Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No